CLINICAL TRIAL: NCT03570593
Title: Evaluation of Early Removal of Urinary Catheter After Radical Surgery for Cervical Cancer Treatment
Brief Title: Removal of Urinary Catheter After Radical Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ricardo dos Reis, Principal Investigator, Barretos Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Barretos Cancer Hospital
Record Dates: First submitted 2018-06-05; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Cervical Cancer; Radical Hysterectomy; Bladder Dysfunction
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrospective Group (No Intervention)
- Prospective Group (Experimental)
  Interventions: Procedure: REMOVAL OF URINARY CATHETER AFTER RADICAL SURGERY

INTERVENTIONS:
Procedure: REMOVAL OF URINARY CATHETER AFTER RADICAL SURGERY — Removal of urinary catheter on the first day after radical surgery
  Arms: Prospective Group

SUMMARY:
Currently, the treatment of cervical cancer in early stages is performed with a radical surgery called Radical Hysterectomy with Pelvic Lymphadenectomy. This surgery, when indicated correctly, in early stages of this disease, has a cure rate of approximately 90% at 5 years, compared to the same Pelvic Radiotherapy. However, it is known that most patients with early stage cervical cancer are young (average age 45) and treating these patients with radiotherapy would have a loss of hormonal function by damage to the ovaries and damage in sexual function by radiotherapy effects in the vagina. Furthermore, if the patient has a pelvic recurrence, the option of radiotherapy treatment could not be offered. Due to the factors listed above, nowadays, in young patients with good clinical conditions and tumors in early stages, radical surgery is a good option. In this radical surgery there is a need for removal of the parametrium, and different degrees of pelvic denervation may occur causing damage of urinary function.Currently, there is no consensus about the correct moment of catheter removal and evaluation of urinary function using the residual urine test. While in some services the urinary catheter is removed on day 1 postoperatively, in others it is removed on the 14th day postoperatively. For these reasons, this study aims to compare the early catheter removal (day 1 postoperatively) versus standard in the investigator's service (7 days postoperatively) withdrawal. If this study detect that the patients may remove the urinary catheter on day 1 postoperatively, much less cost, discomfort, pain and comorbidities associated with the use of indwelling catheter for prolonged periods occur, such as urinary tract infection, use of antibiotics and even hospitalization for this reason.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for this study are women with invasive cervical neoplasia treated with hysterectomy or radical trachelectomy

Exclusion Criteria:

* Patients treated at another cancer service.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2016-07-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Urinary retention | up to 7 days after the surgery
  Measure the urinary retention after the surgery passing an urinary catheter after patient voiding to check the urinary residual

IPD SHARING:
Plan to Share IPD: No